CLINICAL TRIAL: NCT06084572
Title: Prospective Evaluation of PH-impedance Tracings According to the Wingate Consensus, and Influence on Gastro-oesophageal Reflux Disease (GERD) Classification According to the Lyon Consensus.
Brief Title: Prospective Evaluation of PH-impedance Tracings According to the Wingate Consensus, and Influence on GERD Classification According to the Lyon Consensus
Acronym: WinPro
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: WinPro
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: GERD
Keywords: GERD; pH-impedance; Wingate-consensus; Lyon consensus
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GERD patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — FSSG & BEDQ

SUMMARY:
Commonly, in clinical practice an automated analysis of pH-MII tracings is obtained.

DETAILED DESCRIPTION:
All pH-MII performed in UZ Brussel are already reviewed manually according to the Wingate con-sensus and interpreted according to the Lyon consensus. In this study, we will prospectively categorise the reasons for discarding reflux episodes identified by automated analysis during the manual review according to the Wingate consensus, as well as the impact on different parameters related to the interpretation of pH-MII. Based on comments received to our retrospective study, we will evaluate possible confounders to the interpretation, including the indication for referral for pH-MII, symptom severity, use of PPI during pH-MII.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 - 80 years old;
* pH-MII performed off PPI

Exclusion Criteria:

* Prior upper GI endoscopy indicative of structural disease (except for oesophagitis or hiatal hernia).
* Incomplete pH-MII (less than 21 hours recording);
* Ph-MII performed on PPI
* Suboptimal quality of the tracings preventing interpretation in clinical practice;
* Prior oesophageal (including anti-reflux intervention) or gastric surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for pH-MII are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Statistical difference in the GERD categorisation | During baseline visit
  the statistical difference in the distribution of GERD categorisation between automated vs. manual review of the pH-MII tracings

SECONDARY OUTCOMES:
The analysis of the influence of different parameters on application of the Wingate criteria: including the Indication for referral with further classification into predominant oesophageal and extra-oesophageal symptoms; | During baseline visit
The analysis of the influence of different parameters on application of the Wingate criteria: including the GERD Symptom Severity; | During baseline visit
The analysis of the influence of different parameters on application of the Wingate criteria: including the patient being on or off PPI; | During baseline visit
The analysis of the influence of different parameters on application of the Wingate criteria: including MNBI (obtained by automated analysis or manually calculated); | During baseline visit
Presence of significant correlations between censored episodes and pH-MII parameters | During baseline visit
  Correlations including:
  * Acid exposure time;
  * Total number of reflux episodes identified by impedance monitoring;
  * MNBI;
  * PSPWI.
Impact of the Wingate criteria on The number of PSPW; | During baseline visit
Impact of the Wingate criteria on The number of symptoms associated with an impedance episode. | During baseline visit
Impact of the Wingate criteria on the number of impedance episodes with or without acidic reflux | During baseline visit

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - H.U.B, Anderlecht
  - UZ Brussel, Jette
- Technische Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: No